CLINICAL TRIAL: NCT02861170
Title: Effects of a Peri-operative Brief Mindfulness-based Intervention on Post-operative Pain and Disability Among Anxious Patients With Chronic Pain Undergoing Total Hip Arthroplasty - a Feasibility and Acceptability Pilot Randomized Controlled Trial
Brief Title: Effects of a Peri-operative Brief Mindfulness-based Intervention on Post-operative Pain and Disability
Acronym: CALM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was a pilot and after recruitment started it was determined to not be feasible. Therefore study protocol will be reviewed to adjust for changes.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20160105-01H
Record Dates: First submitted 2016-06-23; First posted 2016-08-10 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Chronic Hip Pain; Worries; Pain or Disability; Quality of Life
Keywords: Mindfulness; Chronic Pain; Chronic Hip Pain; Total Hip Arthroplasty; Disability; Quality of Life
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Whole Body Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Mindfulness-Based Intervention (Experimental): Participants in this arm will be provided with an educational brochure and links to videos containing strategies for coping with pain and anxiety as well as a 10-minute mindfulness-based intervention called a body scan at 3 different time-points (T1 - 1 week prior to surgery, T2 - within 4 hours before surgery, and T3 - approximately 24 hours after transfer from recovery to the orthopedic floor).
  Interventions: Behavioral: Brief Mindfulness-Based Intervention
- Education (No Intervention): Participants in this arm will be provided with an educational brochure and links to videos containing strategies for coping with pain and anxiety.

INTERVENTIONS:
Behavioral: Brief Mindfulness-Based Intervention — In addition to the educational materials that will be provided to all participants, the participants in the intervention group will also receive a 10-minute mindfulness-based intervention called a body scan. The body scan is a guided meditation exercise where participants are lead through focusing their attention on their body while maintaining awareness and acceptance of their sensations, emotions, and thoughts without trying to control or change them. The goal of the intervention is to increase mindfulness (i.e., moment-to-moment, non-judgmental and non-reactive awareness of sensations, emotions and thoughts), to provide self-regulation strategies, and to promote healthy and adaptive responses to stress.
  Other Names: Body Scan; Guided Meditation
  Arms: Brief Mindfulness-Based Intervention

SUMMARY:
This study evaluates the effectiveness of a brief mindfulness-based intervention on post-operative pain and disability among anxious patients with chronic pain undergoing total hip arthroplasty.

All participants will receive an educational brochure and links to videos containing strategies for coping with pain and anxiety. The half of the participants who are allocated to the treatment arm will also receive a 10 minute mindfulness intervention called a body scan.

DETAILED DESCRIPTION:
Psychological distress or anxiety is common in patients awaiting surgical procedures and can have impact on both physical and mental health, leading to significantly reduced quality of life. It has been associated with a slower and more complicated postoperative recovery and has been established as an independent predictor of pain and pain related outcomes after surgery.

Pharmacological interventions and provision of information about surgical processes are two ways that pre-operative anxiety is currently addressed. Mindfulness-based interventions have shown positive results in reducing psychological distress and improving pain related outcomes and may be a promising treatment avenue to evaluate in a surgical population.

With the goal of conducting a full-scale definitive trial to investigate the effectiveness of a brief mindfulness-based intervention on post-operative pain and disability among anxious patients with chronic pain undergoing total hip arthroplasty, this pilot study has been developed to demonstrate proof of concept, test/refine the intervention, recruitment, and data collection procedures, and test the intervention's acceptability in the peri-operative setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+) patients presenting at the Pre-Admission Unit (PAU) at the General campus of The Ottawa Hospital (TOH) for total hip arthroplasty (THA)
* History of pain for ≥3 months (chronic pain)
* Anxiety scores of ≥8 on the Generalized Anxiety Disorder 7-item (GAD-7) scale
* Ability to understand oral and written English or French

Exclusion Criteria:

* Refusal or inability to provide consent
* Severe depressive symptoms as indicated by score ≥ 20 on the Patient Health Questionnaire (PHQ-9) scale
* Prior mindfulness training experience
* Pre-planned same day discharge after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale, at approximately 48 hours post-surgery. | Within 4 hours before surgery and approximately 48 hours after transfer from recovery to the orthopedic floor
  The primary outcome will be the mean score of the Brief Pain Inventory (BPI) Interference Scale 48 hours post-surgery. The interference scale measures the degree to which pain interferes in the lives of participants in 7 domains: general activity, mood, walking ability, normal work, relations with other persons, sleep and enjoyment of life on a scale from 0 to 10. The higher the score, the greater the pain interferes with patient's activities.

SECONDARY OUTCOMES:
Change in pain intensity, as measured by the Brief Pain Inventory. | Within 4 hours before surgery and approximately 48 hours after transfer from recovery to the orthopedic floor.
  The Brief Pain Inventory (BPI) Pain Severity Scale measures the severity of pain one feels at worst, at least, on average, and at the time of questionnaire completion on a scale from 0 to 10. The higher the score, the greater the pain severity.
Change in pain catastrophizing, as measured by the Pain Catastrophizing Scale | Within 4 hours before surgery and approximately 48 hours after transfer from recovery to the orthopedic floor.
  The Pain Catastrophizing Scale (PCS) is a 13-item instrument which will evaluate the degree to which patients have negative self-statements and catastrophizing thoughts and ideations when in pain. The PCS uses a 5-point likert scale (0=not at all, 4=all the time) and consists of three subscales (rumination, magnification, helplessness).
Change in mindfulness, as measured by the Short Form Five Facet Mindfulness Questionnaire. | Within 4 hours before surgery and approximately 48 hours after transfer from recovery to the orthopedic floor.
  Mindfulness will be measured using the Short Form Five Facet Mindfulness Questionnaire (FFMQ-SF). The FFMQ-SF is a 24-item instrument measuring five aspects of mindfulness: Non-reactivity to inner experience, observing, describing, acting with awareness, and non-judging of experience. Participants are asked to use a 5-point Likert-type scale (1 = never or rarely true; 5 = very often or always true) to rate how true of them they believe each statement to be.
Change in quality of life, as measured by the EuroQOL-5D | Within 4 hours before surgery and approximately 48 hours after transfer from recovery to the orthopedic floor.
  The EuroQOL-5D (EQ-5D) is a simple-to-use, valid, and sensitive instrument measuring quality of life. It covers 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, or severe problems and participants use a tick box to select the statement that is most representative of their conditions. Participants are also asked to rate, using a visual analogue scale (0 to 100), their state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Poulin, PhD C. Psych, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No